CLINICAL TRIAL: NCT02820961
Title: A Phase 1, Two-Cohort, Open-Label, Drug-Drug Interaction Study of Entinostat and Exemestane in Postmenopausal Women With Locally Recurrent or Metastatic ER+ Breast Cancer
Brief Title: Drug-Drug Interaction Study of Entinostat and Exemestane in Postmenopausal Women With ER+ Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-275-0130
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer; Estrogen Receptor Positive Breast Cancer
Keywords: Breast Neoplasms; Breast Diseases; Exemestane; Protein Kinase Inhibitors; Aromatase Inhibitors; entinostat; Cancer of the Breast; Metastatic Breast Cancer; Hormone Receptor Positive Breast Cancer; Estrogen Receptor; ER+ Breast Cancer; Breast Tumor
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — entinostat; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Active Comparator): Cohort 1 will evaluate exemestane's effect on the PK of entinostat. Each treatment cycle is 28 days.
  Interventions: Drug: entinostat; Drug: exemestane
- Cohort 2 (Active Comparator): Cohort 2 will enroll when Cohort 1 enrollment is complete. Cohort 2 will evaluate entinostat's effect on the PK of exemestane. Each treatment cycle is 28 days.
  Interventions: Drug: entinostat; Drug: exemestane

INTERVENTIONS:
Drug: entinostat — An orally available histone deacetylases inhibitor (HDAC)
  Other Names: SNDX-275; MS-275
Drug: exemestane — Aromatase inhibitor
  Other Names: Aromasin; FCE-24304

SUMMARY:
The purpose of this study is to determine the effect of exemestane on the pharmacokinetics (PK) of entinostat and to determine the effect of entinostat on the PK of exemestane in patients with locally recurrent or metastatic estrogen receptor positive (ER+) breast cancer. Additionally, this study will evaluate the safety and tolerability of entinostat in combination with exemestane, and assess the effectiveness of entinostat in combination with exemestane in terms of best overall response and overall survival.

DETAILED DESCRIPTION:
SNDX-275-0130 is a Phase 1, two-cohort, open-label, drug-drug interaction study of entinostat and exemestane. All patients will be enrolled into one of two cohorts to receive either entinostat monotherapy followed by entinostat plus exemestane (Cohort 1), or exemestane monotherapy followed by exemestane plus entinostat (Cohort 2).

The cohorts will enroll sequentially, meaning that Cohort 1 will enroll prior to Cohort 2. Cohort 1 will evaluate exemestane's effect on the PK of entinostat. Cohort 2 will evaluate entinostat's effect on the PK of exemestane. In both Cohorts, each treatment cycle will be 28 days. Patients will participate in only one cohort.

All patients will be assessed at Screening and at specified times during the conduct of the study using standard clinical and laboratory assessment. Patients will also be assessed for tumor response per standard of care after the Screening Period. Response to treatment will be assessed by computerized tomography (CT), magnetic resonance imaging (MRI) and bone scans as appropriate. Patients will continue receiving their appropriate cycles of study treatment until tumor progression or adverse events (AEs) occur which necessitate discontinuing therapy as determined by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female patients
* Histologically or cytologically confirmed ER+ breast cancer at initial diagnosis and have locally recurrent or metastatic disease that has progressed to where the patient is a candidate to receive exemestane as determined by the Investigator
* Patients receiving palliative radiation at the non-target lesions must be clinically stable prior to receiving the first dose of study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patient must have acceptable, applicable laboratory requirements
* Patients may have a history of brain metastasis provided certain protocol criteria are met
* Able to understand and give written informed consent and comply with study procedures

Exclusion Criteria:

* Rapidly progressive or life-threatening metastases
* Inability to swallow oral medications or gastrointestinal (GI) malabsorption syndromes
* History of significant GI surgery as determined by Investigator
* A medical condition that precludes adequate study treatment or increases patient risk
* Currently enrolled in (or completed within 30 days prior to study drug administration) another investigational drug study

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Cmax, maximum plasma concentration | Approximately 1 year
Tmax, time at which maximum plasma concentration was observed | Approximately 1 year
AUC0-t, area under the plasma concentration-time curve from time zero to the last measurable concentration | Approximately 1 year
AUC0-inf, area under the plasma concentration-time curve from time zero extrapolated to infinity | Approximately 1 year
T1/2, elimination half-life | Approximately 1 year
lambda z , apparent terminal phase elimination constant (λz) | Approximately 1 year
AUC0-τ where τ=168 hours for entinostat and τ=24 hours for exemestane | Approximately 1 year
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), AEs resulting in the permanent discontinuation of study drug, and deaths occurring within 30-days of the last dose of study drug | Approximately 1 year
Changes from baseline in laboratory, vital signs, and electrocardiogram (ECG) values | Approximately 1 year

SECONDARY OUTCOMES:
Best overall tumor response | Approximately 2 years
Overall survival | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Meyers, MD, PhD, Study Director — Syndax Pharmaceuticals
Locations (3):
- United States (3):
  - Sarah Cannon Research Institute HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No